CLINICAL TRIAL: NCT03422146
Title: Antimicrobial and Clinical Efficacy of Cliradex® as Compared With I-Lid'n Lash® Hygiene in Treating Blepharitis: A Randomized, Outcomes-Assessor Masked, Clinical Trial
Brief Title: Antimicrobial and Clinical Efficacy of Cliradex® as Compared With I-Lid'n Lash® Hygiene in Treating Blepharitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P20130792-01H
Record Dates: First submitted 2017-12-12; First posted 2018-02-05 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Blepharitis; Meibomian Gland Dysfunction
MeSH Terms: conditions — Blepharitis; Meibomian Gland Dysfunction | interventions — Tea Tree Oil

STUDY DESIGN:
Intervention Model Description: This study is a single-centre, randomized, outcomes-assessor masked trial with two groups. Patients with chronic blepharitis will be randomized into either the Cliradex® eyelid hygiene or I-Lid 'n Lash® Hygiene group.
  There will be 20 participants enrolled in each group. Although both eyes will receive treatment, only the worse eye will be enrolled in the study. In addition to randomizing the participants into treatment group they will also be placed by chance into either the 3 visit or 4 visit group (n=10 per group).
Who Masked: Investigator, Outcomes Assessor
Masking Description: * Information concerning the group the patient was randomized into will not be available to the physicians that will see the participants at future appointments and grade their outcomes (masked assessor).
  * All microbiology readers will be masked to treatment group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cliradex® eyelid hygiene (Experimental): Cliradex® is a novel over-the-counter eyelid wipe which contains the most active ingredient of TTO. Previous studies have shown the clinical and antimicrobial efficacy of eyelid hygiene with tea tree oil (TTO) in resolving chronic blepharitis.
  Interventions: Other: Tea Tree Oil (TTO)
- I-Lid 'n Lash® Hygiene (Other): Lid 'n Lash® Hygiene, is an over-the-counter eyelid wipe, without any medicinal ingredients,
  Interventions: Other: I-Lid'n Lash® Hygiene

INTERVENTIONS:
Other: Tea Tree Oil (TTO) — Participants will use the Cliradex® eyelid hygiene lid wipe / towelette for BID for 2 weeks
  Arms: Cliradex® eyelid hygiene
Other: I-Lid'n Lash® Hygiene — Patients will use the I-Lid'n Lash® Hygiene lid wipe / towelette for BID for 2 weeks
  Arms: I-Lid 'n Lash® Hygiene

SUMMARY:
Previous studies have shown the clinical and antimicrobial efficacy of eyelid hygiene with tea tree oil (TTO) in resolving chronic blepharitis. Cliradex® is a novel over-the-counter eyelid wipe which contains the most active ingredient of TTO. The present study is a single-centre, randomized, trial comparing Cliradex® eyelid hygiene and I-Lid 'n Lash® Hygiene, another over-the-counter eyelid wipe, without any medicinal ingredients, in treating chronic blepharitis. The Primary Outcome Measure will be the difference in change in the number of CFU's after 2 weeks treatment, between the groups. The Secondary Outcome Measure will be the difference in change in objective clinical signs and symptoms by performing a vision check, a questionnaire, and visual grading, of each participants' blepharitis after 2 weeks treatment, between the groups. The Tertiary Outcome Measures will be the difference in change in microbial CFUs and clinical signs and symptoms between the groups at the 4 and 6 week point, (2 and 4 weeks after discontinuing treatment), to evaluate if the treatment will produce a lasting effect.

Participants will be randomized into one of the treatment arms. They will use the appropriate treatment for two weeks. They will then be re-assessed. They will discontinue treatment at this time, and four weeks later, will be assessed one last time, to see if the temporary treatment provides a lasting effect. A sub-group of ten patients per group will also be randomized to an extra visit. This group will be assessed after two weeks of having stopped the wipes. The same testing and procedures will be performed at this appointment.

DETAILED DESCRIPTION:
Previous studies have shown the clinical and antimicrobial efficacy of eyelid hygiene with tea tree oil (TTO) in resolving chronic blepharitis. This randomized, outcomes-assessor masked, clinical trial aims to determine the efficacy of Cliradex®, which contains the most active ingredient of (TTO), as compared with I-Lid 'n Lash® Hygiene, in treating chronic blepharitis

Blepharitis is a family of inflammatory disease processes of the eyelid. It can be divided anatomically into anterior and posterior blepharitis. Anterior blepharitis refers to inflammation mainly centered around the eyelashes and follicles, while the posterior variant involves the meibomian gland orifices. Anterior blepharitis usually is subdivided further into staphylococcal and seborrheic variants. Frequently, a considerable overlap exists in these processes in individual patients. Blepharitis often is associated with systemic diseases, such as rosacea and seborrheic dermatitis, as well as ocular diseases, such as dry eye syndromes, chalazion, trichiasis, conjunctivitis, and keratitis.1-3

The pathophysiology of blepharitis involves bacterial colonization of the eyelids. This results in direct microbial invasion of tissues, immune system-mediated damage, or damage caused by the production of bacterial toxins, waste products, and enzymes. Colonization of the lid margin is in-creased in the presence of seborrheic dermatitis or meibomian gland dysfunction.1-3

Blepharitis can be difficult to manage because it is often chronic or tends to recur. Despite the cause, eyelid hygiene is the cornerstone of treatment for most cases of blepharitis. This includes the use of commercially available over-the-counter lid cleansing wipes. Previous studies have shown the clinical and microbial efficacy of lid scrubs with tea tree oil (TTO) in resolving chronic blepharitis; however, lid scrubs based on TTO are not convenient for self-administration and cause irritation in some patients.4-11

Cliradex® (Bio-Tissue, Miami, FL) is a commercially available cosmetic pad containing the most active ingredient of TTO, which also exerts potent anti-microbial effects which may eliminate the need for systemic and/or topical antibiotic therapy for blepharitis.

In this trial, the investigators propose to conduct a randomized, outcomes assessor masked, clinical trial to determine the clinical and antimicrobial efficacy of Cliradex® and I-Lid 'n Lash® Hygiene, in improving the signs and symptoms of blepharitis, as well as decreasing the microbial flora in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic blepharitis for duration of at least 3 months.
* Male and female age range: > 18 years old.
* All ethnic groups comparable with the local community.
* Patients able and willing to cooperate with the investigational plan.
* Patients able and willing to complete all postoperative follow-up visits.
* Able to understand and willing to sign a written informed consent.

Exclusion Criteria:

* Patients who are currently engaged in another clinical trial.
* Patients who are unwilling or unable to give consent.
* Patients who are unwilling to accept randomization.
* Patients who will not be able to return for scheduled visits.
* Children under 18.
* Concomitant use of ophthalmic topical medications (excluding non-preserved tear substitutes).
* Concomitant use of systemic antibiotics or steroids.
* Active ocular infection or allergy.
* Previous surgery on the eyelids such as blepharoplasty.
* Abraded skin on or around the eyelids.
* Patients unable to close eyes or uncontrolled blinking.
* Previous allergic reaction to TTO-containing products or cosmetic fragrance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-02-19 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Evidence of microbiologic improvement | 2 weeks
  difference in change in the number of CFU's after 2 weeks treatment, between the groups. (Note: colony counts over 200 will not be counted but reported as >200)

SECONDARY OUTCOMES:
Improvement in signs & symptoms of blepharitis based on visual grading scale | 2 weeks
  The Secondary Outcome Measure will be the difference in change in objective clinical signs and symptoms using a visual grading scale
Improvement in signs & symptoms of blepharitis based on participant questionnaire | 2 weeks
  The Secondary Outcome Measure will be the difference in change in objective clinical signs and symptoms using a questionnaire after 2 weeks treatment between the groups.

OTHER OUTCOMES:
Evidence of continued microbiologic improvement after discontinuing blepharitis treatment | 2 & 4 weeks post discontinuation of treatment
  difference in change in the number of CFU's at 2 & 4 weeks post discontinuation of treatment, between the groups. (Note: colony counts over 200 will not be counted but reported as >200)
Evidence of continued improvement in signs & symptoms of blepharitis, based on grading scale, after discontinuing blepharitis treatment | 2 & 4 weeks post discontinuation of treatment
  The Outcome Measure will be the difference in change in objective clinical signs and symptoms using a visual grading scale
Evidence of continued improvement in signs & symptoms of blepharitis, based on participant questionnaire, after discontinuing blepharitis treatment | 2 & 4 weeks post discontinuation of treatment
  The Outcome Measure will be the difference in change in objective clinical signs and symptoms using a questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Setareh Ziai, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Health Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No